CLINICAL TRIAL: NCT01278576
Title: An Efficacy Comparison of Botulinum Toxin A Injection Into Two Different Sites in Gastrocnemius Muscle for the Treatment of Spastic Patients, Randomized Controlled Trial
Brief Title: Botulinum Toxin A Adult Gastrocnemius Muscle Study
Acronym: BTX-A
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Collaborators: Bobath Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sun Im, Assistant Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCMC10AH07
Record Dates: First submitted 2011-01-10; First posted 2011-01-19 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2011-01

CONDITIONS: Muscle Spasticity; Stroke
Keywords: Muscle spasticity; Stroke; Botulinum Toxins; Lower extremity; Ankle
MeSH Terms: conditions — Muscle Spasticity; Stroke | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intramuscular ending Targeting (Experimental): Botox 200 units placed at the upper 2/10-3/10 length of the GCM
  Interventions: Drug: BOTOX-A®
- Midbelly Targeting (Active Comparator): A total of 200 units will be placed at the four quadrants of the midbelly portion of the GCM.
  Interventions: Drug: BOTOX-A®

INTERVENTIONS:
Drug: BOTOX-A® — 200 units, single treatment only
  Other Names: Generic Name: Botulinum toxin type A

SUMMARY:
The study aims to compare the effectiveness of BOTOX-A® (botulinun toxin A) placed between two different injection sites, namely at the proximal portion of the gastrocnemius(GCM) versus at the midbelly of the GCM.

DETAILED DESCRIPTION:
Previous studies have used the midbelly of a muscle as the position where the motor endplates are most densely located. The reasoning behind this method was based on the previous works that showed most bands of cholinesterase activity to be located in specific topographical patterns at the center of the muscle fiber. These results have been used as landmarks to place the injections. Current standard guidelines recommend that botulinum toxin be placed at the 4 quadrants of the midbelly portion of the gastrocnemius (GCM) muscle. However, recent cadaveric research studies on the distribution of the intramuscular endings of the GCM suggest that the highest branch density is found within the upper 20-30% length of the calf. Therefore, in accordance to the theory that effect of botulinum toxin are greatest at sites where the intramuscular endings are most dense, the location where these toxins should be placed would be at these proximal sites of the GCM rather than at the midbelly.

40 recruited patients will be allocated into either the intramuscular ending targeted (ie.upper portion of calf) or midbelly targeted group.

Each subject will undergo a total number of 4 assessments; prior to the injection and 2,4and 8 weeks post injection.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 20 < age < 70 year old
* Hemiplegia documented after ischemic or hemorrhagic stroke, documented by CT (computed tomography) or MRI (magnetic resonance imaging) scan
* Time between the onset of stroke < 24 months
* Individuals who have been medically stable for at least 4 weeks prior to study enrollment
* Confirmed equinovarus with spastic hypertonia of the ankle
* Spasticity as defined by a MAS greater than grade 1 +
* Botulinum toxin -naive patients
* Participants who can complete the 10 meter walking test with caregiver or walking tool assistance within 8 and 45 seconds, on 2 occasions
* Participants who will have stable treatment regimen and concomitant medication during the trial period

Exclusion Criteria:

* The patient has any of the following medical conditions that is contraindication to botulinum toxin exposure; pregnancy, lactation, neuromuscular disease, aminoglycoside, antibiotic concurrent to botulinum toxin treatment
* Fixed contracture of the ankle, previous history of surgical procedure performed on the ankle
* Cognitive deficit that disables patients to give informed consent to the procedure
* Concomitant progression of any CNS (central nervous system) or PNS (peripheral nervous system), or myopathy, or uncontrolled seizure. Underlying CNS insult should be controlled and in stable condition with no further risk of progression and further deterioration of patient's current neurological status. Those with multiple sclerosis or multiple systemic atrophy are to be excluded
* Significant cutaneous or joint inflammation
* URI or other systemic infection that would mandate the use of antibiotic concurrent to botulinum toxin injection
* Anticoagulation treatment with INR (International Normalized Ratio) greater than 3.0
* Upper extremity spasticity greater than MAS grade 4 that may limit gait function
* Subjects with previous episodes of motor point block injection using phenol or other chemodenervating agents
* Subjects with intrathecal baclofen pump

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline for EMG (electromyogram) activity | week 8
  Surface EMG

SECONDARY OUTCOMES:
Change from baseline of GCM tone a measured on the Modified Ashworth Scale (MAS) | Change from baseline at 8 weeks
Change from baseline of Ankle Range of motion | Change from baseline at 8 weeks
  Passive range of motion of the ankle at resting state with the use of goniometer
Change from baseline of gait speed with 10 meters walk test | Change from baseline at 8 weeks
  Change from baseline at 8 weeks
Change from baseline of ABILOCO scale | Change from baseline at 8 weeks
Change from baseline of Disability Assessment Scale | Change from baseline at 8 weeks
Change from baseline of Functional Ambulation Category Scale | Change from baseline at 8 weeks
Change of baseline of Lindmark Modified Fugyl Meyer Scale | Change from baseline at 8 weeks
Change from baseline of Tardieu angle of ankle | Change from baseline at 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sun Im, MD, PhD, Principal Investigator — Department of Rehabilitation Medicine, Bucheon St Mary's Hospital, Catholic University of Korea, College of Medicine
Locations (2):
- South Korea (2):
  - Department of Rehabilitation Medicine Bucheon St Mary's Hospital, Catholic University of Korea, College of Medicine, Bucheon-si, Kyounggido
  - Bobath Memorial Hospital, Songnam, Kyoungido